CLINICAL TRIAL: NCT01664260
Title: Elucidation of Efficacy Mechanism of N-acetylcysteine in Patients With Posttraumatic Stress Disorder: An 8-week Multimodal Neuroimaging and Neurocognitive Study
Brief Title: Efficacy Mechanism of N-acetylcysteine in Patients With Posttraumatic Stress Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The research project has been cancelled before any participants were enrolled.
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iklnac
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; N-acetylcysteine; Magnetic Resonance Imaging
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine + Escitalopram (Experimental): The subjects with posttraumatic stress disorder, treated with N-acetylcysteine in addition to escitalopram
  Interventions: Drug: N-acetylcysteine
- Placebo + Escitalopram (Placebo Comparator): The subjects with posttraumatic stress disorder, treated with placebo in addition to escitalopram
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — 0 - 8 week: 10 mg escitalopram a day + 1200 mg N-acetylcysteine twice a day
  Arms: N-acetylcysteine + Escitalopram
Drug: Placebo — 0 - 8 week: 10 mg escitalopram a day + 1200 mg Placebo twice a day
  Arms: Placebo + Escitalopram

SUMMARY:
It has been suggested that N-acetylcysteine exerts neuroprotective effects by regulating neurotransmitters and cell signaling pathways. We hypothesize that oral N-acetylcysteine augmentation will help reduce symptoms in patients with posttraumatic stress disorder as well as improve cognitive functions. We also expect that the N-acetylcysteine augmentation will induce change in structural, functional, and neurochemical aspects of the brain.

In this study, we plan to conduct a randomized, double-blind, placebo-controlled augmentation study with N-acetylcysteine in addition to escitalopram. We will assess the efficacy and safety of the N-acetylcysteine augmentation.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 year-old male or female
* Posttraumatic stress disorder diagnosed by SCID-IV
* Written informed consent

Exclusion Criteria:

* Medication treatment for posttraumatic stress disorder within 2 weeks
* Neurologic disease (eg., penetrating or open head injury, epilepsy, multiple sclerosis, brain tumor, cerebrovascular diseases)
* Any other axis I psychiatric disorder
* IQ below 80
* Contraindications to magnetic resosnance imaging (e.g., pacemaker implantation, claustrophobia, etc.)
* Any psychotropic medication within 2 weeks
* Unstable medical illness or severe abnormality in laboratory test at screening assessment
* Women who are pregnant, breastfeeding, or planning pregnancy
* History of myocardial infarction within 6 months
* Current diagnosis of duodenal ulcer or asthma
* Contraindications to drugs used in the study (e.g., epilepsy, uncontrolled narrow-angle glaucoma, etc.)
* Allergy or intolerance to the study drug

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11-01 (Estimated); Primary Completion 2016-12-01 (Estimated); Study Completion 2016-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in brain structure, function, and biochemical metabolism, analyzed using the computational approach | Baseline, 8th weeks
Change from baseline in Clinician-administered PTSD scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Clinician-administered PTSD scale scores at 8th weeks | Baseline, 8th weeks

SECONDARY OUTCOMES:
Change from baseline in Hamilton depression rating scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Hamilton depression rating scale scores at 8th weeks | Baseline, 8th weeks
Change from baseline in Hamilton anxiety rating scale scores at 4th weeks | Baseline, 4th weeks
Change from baseline in Hamilton anxiety rating scale scores at 8th weeks | Baseline, 8th weeks
Number of participants with adverse events | 4th weeks
Number of participants with adverse events | 8th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inkyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University Medical Center, Seoul, South Korea